CLINICAL TRIAL: NCT04591691
Title: Predictive and Diagnostic Biomarkers for Diabetic Foot Ulcers - C-myc and Phosphorylated Glucocorticoid Receptor
Brief Title: C-myc Biomarker Study for Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Indiana University (Other); Stanford University (Other); University of Miami (Other); University of Pittsburgh (Other); University of California, San Francisco (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Cathie Spino, ScD, Research Professor of Biostatistics, SABER Director, University of Michigan
Other Study IDs: HUM00168547; 1U24DK122927-01 (NIH)
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Diabetes; Diabetic Foot; Diabetic Foot Ulcer; Diabetic Wound
Keywords: biomarker; C-myc; phosphorylated glucocorticoid receptor; DFC; Diabetic Foot Consortium
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Wound edge issue specimens are collected from the wound edge at Week 0 and, if clinically indicated, at Week 4 of the study. Investigators sample full thickness skin of a wound edge that includes epidermis and dermis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center observational cohort study of patients with diabetic foot ulcers (DFU) to develop and validate potential tissue-based biomarkers that predict complete wound healing. Eligible and consented participants will begin standard of care treatment after collection of tissue specimens from the wound's edge. An additional tissue specimen is collected at 4 weeks if clinically indicated. Tissues will be tested for c-myc and phosphorylated glucocorticoid receptor (p-GR) levels using validated protocols at a central laboratory. Participants will be followed weekly for up to 12 weeks or until complete wound healing (whichever occurs first). One final assessment 2 weeks after complete wound healing will occur to confirm healing.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or older.
4. Clinically diagnosed with diabetes or meeting the American Diabetes Association (ADA) criteria.
5. Foot ulcer of diabetic etiology, with all of the following characteristics:

   1. Ulcer size > 0.5 cm2 and < 12 cm2 at least 2 cm from any other ulcer, and
   2. Ulcer with Wagner grade 1 or 2 In case of multiple ulcers, select the largest ulcer that meets inclusion criteria.
6. Patients with neuropathic or neuro-ischemic ulcers with adequate circulation to allow healing to the affected extremity as demonstrated by at least 2 of the following within 6 months of Visit 1:

   1. Ankle brachial index (ABI) ≥ 0.6 with Doppler Waveforms, or
   2. Absolute ankle pressure ≥ 70 mm Hg, or
   3. Toe pressure ≥ 40 mmHg, or
   4. TcPO2 ≥ 40 mmHg
7. Willingness to comply with standard of care which includes an initial surgical debridement of the wound.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patient participating in an interventional clinical trial within 1 month of Visit 1
2. Currently receiving radiation to target area or chemotherapy
3. Participants with Charcot's foot or other foot deformities that prevents adequate targeted ulcer offloading
4. Participant with active severe infection or osteomyelitis at the time of screening
5. History of cancer within last 3 years, other than non-melanoma skin cancer
6. Known or suspected malignancy of current study ulcer
7. Use of adjunctive therapy within previous 30 days
8. Currently receiving medication considered to be systemic glucocorticoids
9. Plan to perform a vascular intervention, such as surgical bypass, angioplasty or stenting, or < 1 month from a prior ipsilateral vascular intervention
10. Any history of concomitant medical condition that, in the opinion of the investigator(s), would compromise the participant's ability to safely complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Type 1 or Type 2 Diabetic patients with a diabetic foot ulcer
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with complete wound healing by week 12, defined as complete wound closure where there is skin re-epithelialization without drainage or dressing requirements | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marjana Tomic-Canic, Principal Investigator — University of Miami
Locations (6):
- United States (6):
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Miami, Miami, Florida
  - Indiana University Health, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided